CLINICAL TRIAL: NCT03675724
Title: AFFIRM-LITE: A Phase 2 Randomized, Placebo-Controlled Study of Alleviation by Fisetin of Frailty, Inflammation, and Related Measures in Older Adults
Brief Title: Alleviation by Fisetin of Frailty, Inflammation, and Related Measures in Older Adults
Acronym: AFFIRM-LITE
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert J. Pignolo, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-007332
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Frail Elderly Syndrome
Keywords: Frailty; Inflammation; Elderly; Aging
MeSH Terms: conditions — Frailty; Inflammation | interventions — fisetin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Fisetin 20mg/kg/day, orally for 2 consecutive days
  Interventions: Dietary Supplement: Fisetin
- Placebo (Placebo Comparator): Placebo capsules orally for 2 consecutive days
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Dietary Supplement: Fisetin — Flavonoid Family
  Arms: Treatment
Drug: Placebo oral capsule — Placebo
  Arms: Placebo

SUMMARY:
This is a pilot study to test the efficacy of the anti-inflammatory drug (Fisetin) in reducing inflammatory factors in blood in elderly adults and to test the efficacy of the drug (Fisetin) in reducing frailty and markers of inflammation, insulin resistance, and bone resorption in elderly adults.

DETAILED DESCRIPTION:
To the researchers' knowledge, there are no published studies utilizing Fisetin in alteration of frailty markers. Several studies involve use of Fisetin for its anti-oxidative and anti-apoptotic effects in animal models. Fisetin may reduce oxidative stress, alleviate hyperglycemia, and improve kidney function. No one has evaluated the biologic markers of inflammation and frailty in older adults. The researchers plan to evaluate markers of frailty and markers of inflammation, insulin resistance, and bone resorption while maintaining bone formation in older adults.

ELIGIBILITY:
Inclusion Criteria

• Age ≥ 70 years

Exclusion Criteria

* Unable or unwilling to give informed consent
* Pregnant
* Body weight >150 kg or body mass index (BMI) > 50
* QTc>450 msec
* Total bilirubin >2X upper limit of normal
* Inability to tolerate oral medication
* Abnormality in any of the screening laboratory studies (see below)
* Human immunodeficiency virus infection
* Known active hepatitis B or C infection
* Invasive fungal or viral infection
* Known hypersensitivity or allergy to fisetin
* Uncontrolled pleural/pericardial effusions or ascites
* New/active invasive cancer except non-melanoma skin cancers
* Subjects taking medications that are sensitive to substrates or substrates with a narrow therapeutic range for CYP3A4, CYP2C8, CYP2C9, or CYP2D6 or strong inhibitors or inducers of CYP3A4 (e.g. cyclosporine, tacrolimus or sirolimus). If antifungals are absolutely necessary from an infectious disease perspective, then they will be allowed only if the levels are therapeutic.
* Strong inhibitors of CYP3A4. See Appendices 1-3.
* Tyrosine kinase inhibitor therapy
* Known hypersensitivity or allergy to fisetin
* Subjects on quinolone antibiotic therapy for treatment or for prevention of infections within 10 days.
* Subjects taking H2-antagonists and unwilling to discontinue therapy for 1 week before and 2 weeks following enrollment.
* Subjects taking potentially senolytic agents within the last year: Fisetin, Quercetin, Luteolin, Dasatinib, Piperlongumine, or Navitoclax
* Subjects currently taking drugs that induce cellular senescence: alkylating agents, anthracyclines, platins, other chemotherapy
* Subjects taking the following antimicrobial agents: Aminoglycosides, Azole antifungals (fluconazole, miconazole, voriconazole, itraconazole), Macrolides (clarithromycin,erythromycin), Antivirals (nelfinavir, indinavir, saquinavir, ritonavir, elbasvir/grazoprevir), Rifampin
* Subjects taking proton pump inhibitors who are unable or unwilling to reduce or hold therapy 2 days prior to and during the 2-day Fisetin dosing
* Subjects taking the following other drugs if they cannot be held for at least 2 days before and during administration of Fisetin: digoxin, lithium, all statins, repaglidine, bosentan, gemfibrozil, olmesartan, enalapril, valsartan, methotrexate, corticosteroids, , eluxadoline, eltrombopag, nitroglycerin, pioglitazone, glyburide, enzalutamide, ezetimibe, colchicine, imatinib, cyclosporine, tacolimus, sirolimus, carbamazepine, flecainide, phenytoin, phenobarbital, rifampicin, theophylline, celecoxib, desipramine, thioridazine, venlafaxine, tizanidine, atomoxetine, voriconazole, citalopram, diazepam, escitalopram, propranolol, clozapine, cyclobenzaprine, mexiletine, olanzapine, ondansetron, riluzole
* In order to ensure vitamin D sufficiency, we will also exclude subjects with serum 25-hydroxyvitamin D levels of < 20 ng/ml.
* Presence of any condition that the Investigator believes would put the subject at risk or would preclude the patient from successfully completing all aspects of the trial.

Behavioral Modification - Participants will be educated about the risk of excessive caffeine usage. Participants will be encouraged to reduce use by 50% prior to and during the 2-day drug dosing period. Due to drug-drug interaction, subjects may not clear the caffeine from their system properly/as usual.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Decrease in blood inflammation markers | Seven Days
  Percent decrease in blood inflammation markers

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pignolo, MD, PhD, Principal Investigator — Mayo Clinic; Sundeep Khosla, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No